CLINICAL TRIAL: NCT00568529
Title: Phase II Study on Combination of Capecitabine and Oxaliplatin in Patients With Relapsed or Refractory Gastric Cancer
Brief Title: Combination of Capecitabine and Oxaliplatin in Patients With Relapsed or Refractory Gastric Cancer
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: There are not enough patients enrolled.
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University cancer hospital, Fudan University cancer hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XELOX-AGC
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2009-08

CONDITIONS: Gastric Cancer
Keywords: Advanced gastric cancer; Response rate; Side effects; time to progression; overall survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combine Chemotherapy (Experimental): XELOX(Xeloda and oxaliplatin combination)
  Interventions: Drug: Capecitabine and Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine and Oxaliplatin — Capecitabine 1000mg/m2 Bid d1-14 Oxaliplatin 130mg/m2 d1 q3w
  Other Names: XELOX(Xeloda and oxaliplatin combination)

SUMMARY:
The purpose of this study is to evaluate the efficacy and overall survival of the regimen of XELOX (Xeloda and oxaliplatin combination) in the patients with relapsed and refractory gastric cancer.

DETAILED DESCRIPTION:
The result of treatment in relapsed and refractory gastric cancer is still not satisfactory. For the moment, the combination of 5-Fu and cisplatin is regularly used. Capecitabine and Oxaliplatin are new generation drugs of 5-Fu and cisplatin. The current study is to evaluate the efficacy and toxicity of this combination.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Patients with histologically confirmed, unresectable, recurrent and/or metastatic gastric adenocarcinoma
* ECOG performance status ≤1
* Measurable diseases according to the RECIST
* Relapse or refractory after the first-line chemotherapy
* Sign ICF,normal laboratory findings:absolute neutrophil count and platelet count ≥ 2.0×109/L and 80×109/L, respectively, hepatic function (total serum bilirubin ≤ UNL, transaminases ≤ 1.5 times upper normal limit) and renal function (calculated creatinine clearance ≥ 60 ml/min).

Exclusion Criteria:

* Relapse within 6 months after adjuvant chemotherapy which contained oxaliplatin
* Have used any of drugs in the regimen in first-line chemotherapy
* Pregnant or lactating women,serious uncontrolled diseases and intercurrent infection
* The evidence of CNS metastasis
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Received other chemotherapy regimen after metastasis
* Participated in other clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 2-6 months

SECONDARY OUTCOMES:
time to progression and overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China